CLINICAL TRIAL: NCT00870818
Title: An Extension of Study CP-MGA031-01 to Evaluate the Long-Term Efficacy and Safety of Teplizumab (MGA031), a Humanized, FcR Non-Binding, Anti-CD3 Monoclonal Antibody, in Patients With Recent-Onset Type 1 Diabetes Mellitus
Brief Title: Protege Extension Trial - Long Term Follow Up Trial for Subjects Who Completed the Protege Study (CP-MGA031-01)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Business decision
Sponsor: MacroGenics (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: CP-MGA031-02
Record Dates: First submitted 2009-03-26; First posted 2009-03-27 (Estimated); Results first posted 2023-08-09 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-07

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Teplizumab; Protege; MGA031; Monoclonal antibody; Type 1 Diabetes Mellitus; T1DM; MacroGenics
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Blood Specimen Collection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (5):
- Double-blind Herold Regimen (Experimental): Patients who had been assigned to Herold Regimen in Segment 2 of Study CP-MGA031-01 were enrolled to gather additional safety and efficacy data.
  Interventions: Diagnostic Test: Blood samples for safety; Behavioral: Patient reported outcome questionnaires; Diagnostic Test: Analysis of T-cell subsets
- Double-blind 33.3% Herold Regimen (Experimental): Patients who had been assigned to 33.3% Herold Regimen in Segment 2 of Study CP-MGA031-01 were enrolled to gather additional safety and efficacy data.
  Interventions: Diagnostic Test: Blood samples for safety; Behavioral: Patient reported outcome questionnaires; Diagnostic Test: Analysis of T-cell subsets
- Double-blind Curtailed Herold Regimen (Experimental): Patients who had been assigned to Curtailed Herold Regimen in Segment 2 of Study CP-MGA031-01 were enrolled to gather additional safety and efficacy data.
  Interventions: Diagnostic Test: Blood samples for safety; Behavioral: Patient reported outcome questionnaires; Diagnostic Test: Analysis of T-cell subsets
- Double-blind Placebo (Placebo Comparator): Patients who had been assigned to Placebo in Segment 2 of Study CP-MGA031-01 were enrolled to gather additional safety and efficacy data.
  Interventions: Diagnostic Test: Blood samples for safety; Behavioral: Patient reported outcome questionnaires; Diagnostic Test: Analysis of T-cell subsets
- Open-label Herold Regimen (Experimental): Patients who had been assigned to Herold Regimen in Segment 1 of Study CP-MGA031-01 were enrolled to gather additional safety and efficacy data.
  Interventions: Diagnostic Test: Blood samples for safety; Behavioral: Patient reported outcome questionnaires; Diagnostic Test: Analysis of T-cell subsets

INTERVENTIONS:
Diagnostic Test: Blood samples for safety — serum chemistry, hematology, infection screen, thyroid function, Insulin, hemoglobin A1c,and autoantibodies
Behavioral: Patient reported outcome questionnaires — EQ-5D, Peds QL, Low blood sugar survey, and hospitalization information.
Diagnostic Test: Analysis of T-cell subsets — CD3, CD4, CD8, CD19, CD3+ CD16+ CD56+ subsets; CD3-CD16+ CD56+ subsets; CD4+CD25+, CD8+CD25+, CD4+CD69+, CD8+CD69+, CD4+CD40+ subsets CD4+ and CD8+CD25+FoxP3+Treg Subsets

SUMMARY:
The purpose of this study is to assess the long term safety and efficacy in subjects with Type 1 Diabetes Mellitus who completed the Protege Study (CP-MGA031-01).

DETAILED DESCRIPTION:
The primary objective of the extension study is to assess long-term safety, with particular focus on the development of serious adverse events (SAEs), adverse events of special interest (AESIs) including opportunistic infections and lymphoproliferative disease, and other immediately reportable events (IREs), in subjects with recent-onset T1DM who complete CP-MGA031-01.

The secondary objectives of the extension study are to: 1) assess long-term efficacy; 2) evaluate immunological effects(North America only); 3) measure anti-teplizumab antibody levels;4) assess Health Related Quality of Life Questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Complete Protocol CP-MGA031-01 (i.e., all subjects who complete Study Day 728, regardless of how many doses of study drug are received).
2. Provide written informed consent.

Exclusion Criteria:

None

Ages: 10 Years to 37 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 219 (Actual)
Dates: Start 2009-02; Primary Completion 2011-02 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Atlanta Diabetes Associates, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Open-label Herold Regimen | Double-blind Herold Regimen | Double-blind 33.3% Herold Regimen | Double-blind Curtailed Herold Regimen | Double-blind Placebo
Started | 32 | 73 | 38 | 38 | 38
Completed 6 Months | 31 | 22 | 13 | 13 | 11
Completed 12 Months | 27 | 2 | 3 | 2 | 2
Completed 18 Months | 5 | 0 | 0 | 0 | 0
Completed 21 Months | 1 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 32 | 73 | 38 | 38 | 38
Not completed — Lost to Follow-up | 3 | 2 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 2 | 0
Not completed — Terminated by sponsor | 29 | 70 | 36 | 36 | 38
Not completed — Other | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Open-label Herold Regimen | Double-blind Herold Regimen | Double-blind 33.3% Herold Regimen | Double-blind Curtailed Herold Regimen | Double-blind Placebo | Total
Number analyzed (Participants) | 32 | 73 | 38 | 38 | 38 | 219
Age, Continuous [Median (Full Range); unit: years] | 14.0 [10.0 to 34.0] | 18.0 [9.0 to 35.0] | 18.5 [10.0 to 31.0] | 16.0 [8.0 to 32.0] | 16.5 [10.0 to 34.0] | 18.0 [8.0 to 35.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 32 | 12 | 9 | 14 | 74
  Male | 25 | 41 | 26 | 29 | 24 | 145
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 1 | 1 | 0 | 5
  Not Hispanic or Latino | 31 | 71 | 37 | 37 | 38 | 214
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 5 | 27 | 12 | 13 | 15 | 72
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 27 | 45 | 26 | 25 | 23 | 146
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 16 | 19 | 11 | 11 | 8 | 65
  Czechia | 7 | 8 | 4 | 4 | 4 | 27
  India | 5 | 26 | 12 | 13 | 15 | 71
  Romania | 4 | 3 | 1 | 2 | 2 | 12
  Ukraine | 0 | 6 | 4 | 3 | 2 | 15
  Israel | 0 | 4 | 4 | 2 | 4 | 14
  Spain | 0 | 4 | 2 | 1 | 2 | 9
  Estonia | 1 | 1 | 0 | 1 | 1 | 4
  Latvia | 0 | 1 | 0 | 0 | 0 | 1
  Poland | 0 | 1 | 0 | 0 | 0 | 1
  Sweden | 0 | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants Who Experience an Adverse Event, Serious Adverse Event or Adverse Event of Special Interest.
Time Frame: Duration of study participation up to 15 months
Measure: Count of Participants; unit: Participants
Arm/Group | Open-label Herold Regimen | Double-blind Herold Regimen | Double-blind 33.3% Herold Regimen | Double-blind Curtailed Herold Regimen | Double-blind Placebo
Number analyzed (Participants) | 32 | 73 | 38 | 38 | 38
Participants | 8 | 8 | 3 | 10 | 4

2. Secondary Outcome: Proportion of Subjects in Segment 2 With Both a Total Daily Insulin Dose of Less Than 0.5 U/kg/Day and Hemoglobin A1c (HbA1c) Level of Less Than 6.5%.
Time Frame: Month 6
Population: Because the study was terminated early with a limited number of subjects and subject visits, the data are only summarized. Too few data are available for meaningful analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Open-label Herold Regimen | Double-blind Herold Regimen | Double-blind 33.3% Herold Regimen | Double-blind Curtailed Herold Regimen | Double-blind Placebo
Number analyzed (Participants) | 29 | 20 | 10 | 11 | 8
Participants | 3 | 3 | 0 | 1 | 0

3. Secondary Outcome: Proportion of Subjects in Segment 2 With Both a Total Daily Insulin Dose of Less Than 0.5 U/kg/Day and Hemoglobin A1c (HbA1c) Level of Less Than 6.5%.
Time Frame: Month 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Open-label Herold Regimen | Double-blind Herold Regimen | Double-blind 33.3% Herold Regimen | Double-blind Curtailed Herold Regimen | Double-blind Placebo
Number analyzed (Participants) | 26 | 2 | 2 | 2 | 2
Participants | 4 | 1 | 0 | 1 | 0

4. Secondary Outcome: Proportion of Subjects With HbA1c <6.5%
Time Frame: Month 6
Measure: Count of Participants; unit: Participants
Arm/Group | Open-label Herold Regimen | Double-blind Herold Regimen | Double-blind 33.3% Herold Regimen | Double-blind Curtailed Herold Regimen | Double-blind Placebo
Number analyzed (Participants) | 30 | 13 | 13 | 13 | 11
Participants | 5 | 6 | 3 | 2 | 0

5. Secondary Outcome: Mean HbA1c at 6 Months
Time Frame: 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | Open-label Herold Regimen | Double-blind Herold Regimen | Double-blind 33.3% Herold Regimen | Double-blind Curtailed Herold Regimen | Double-blind Placebo
Number analyzed (Participants) | 30 | 22 | 13 | 13 | 11
percentage of glycosylated hemoglobin | 8.24 (2.063) | 8.25 (0.262) | 8.25 (2.709) | 7.83 (1.489) | 8.10 (1.009)

6. Secondary Outcome: Mean HbA1c at 12 Months
Time Frame: Month 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | Open-label Herold Regimen | Double-blind Herold Regimen | Double-blind 33.3% Herold Regimen | Double-blind Curtailed Herold Regimen | Double-blind Placebo
Number analyzed (Participants) | 27 | 2 | 2 | 2 | 2
percentage of glycosylated hemoglobin | 7.81 (2.155) | 6.30 (0.141) | 6.35 (0.354) | 6.05 (0.778) | 6.95 (0.919)

7. Secondary Outcome: C-peptide Area Under the Curve (AUC) at 6 Months
Description: This outcome measure summarizes the mean and standard deviation of the observed value.
Time Frame: Month 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: min*nmol/L
Arm/Group | Open-label Herold Regimen | Double-blind Herold Regimen | Double-blind 33.3% Herold Regimen | Double-blind Curtailed Herold Regimen | Double-blind Placebo
Number analyzed (Participants) | 30 | 22 | 13 | 11 | 10
min*nmol/L | 0.30 (0.195) | 0.45 (0.360) | 0.25 (0.301) | 0.25 (0.248) | 0.37 (0.399)

8. Secondary Outcome: C-peptide AUC at 12 Months
Description: This outcome measure summarizes the mean and standard deviation of the observed value.
Time Frame: Month 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: min*nmol/L
Arm/Group | Open-label Herold Regimen | Double-blind Herold Regimen | Double-blind 33.3% Herold Regimen | Double-blind Curtailed Herold Regimen | Double-blind Placebo
Number analyzed (Participants) | 27 | 2 | 2 | 2 | 2
min*nmol/L | 0.32 (0.183) | 0.56 (0.123) | 0.26 (0.276) | 0.59 (0.036) | 0.19 (0.058)

9. Secondary Outcome: Total Daily Insulin Usage at 6 Months
Time Frame: Month 6
Measure: Mean (Standard Deviation); unit: units/kg/day
Arm/Group | Open-label Herold Regimen | Double-blind Herold Regimen | Double-blind 33.3% Herold Regimen | Double-blind Curtailed Herold Regimen | Double-blind Placebo
Number analyzed (Participants) | 30 | 20 | 10 | 11 | 8
units/kg/day | 0.71 (0.362) | 0.71 (0.451) | 0.64 (0.274) | 0.81 (0.433) | 0.60 (0.251)

10. Secondary Outcome: Total Daily Insulin Usage at 12 Months
Time Frame: Month 12
Measure: Mean (Standard Deviation); unit: units/kg/day
Arm/Group | Open-label Herold Regimen | Double-blind Herold Regimen | Double-blind 33.3% Herold Regimen | Double-blind Curtailed Herold Regimen | Double-blind Placebo
Number analyzed (Participants) | 26 | 2 | 2 | 2 | 2
units/kg/day | 0.67 (0.280) | 0.47 (0.073) | 0.49 (0.076) | 0.40 (0.147) | 0.76 (0.272)

11. Secondary Outcome: Mean Values for Participant-reported Outcomes on the 5-dimension European Quality of Life Questionnaire. (EQ-5D)
Description: The EQ-5D is a self-reported survey that measures quality of life across 5 domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is scored on a 3-level severity ranking that ranges from "no problems", "some problems", and "extreme problems". The lowest possible score is 5 and the highest possible score is 15. Lower scores indicate better quality of life.
Time Frame: Month 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open-label Herold Regimen | Double-blind Herold Regimen | Double-blind 33.3% Herold Regimen | Double-blind Curtailed Herold Regimen | Double-blind Placebo
Number analyzed (Participants) | 27 | 18 | 10 | 11 | 9
units on a scale | 5.3 (0.53) | 5.8 (1.25) | 5.2 (0.63) | 5.1 (0.30) | 5.7 (1.12)

12. Secondary Outcome: Mean Values for Participant-reported Outcomes on the EQ-5D
Description: as for outcome 11
Time Frame: Month 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open-label Herold Regimen | Double-blind Herold Regimen | Double-blind 33.3% Herold Regimen | Double-blind Curtailed Herold Regimen | Double-blind Placebo
Number analyzed (Participants) | 26 | 2 | 2 | 2 | 2
units on a scale | 5.1 (0.33) | 6.52 (2.12) | 5.0 (0.00) | 5.0 (0.00) | 6.0 (1.41)

13. Secondary Outcome: Pediatric Quality of Life Questionnaire Total Score
Description: The 23-item PEDs QL generic core scales were designed to measure the core dimensions of health (physical, emotional, social and school functioning). Answers are scored from 0 meaning never to 4 meaning almost always. Lower scores indicated higher quality of life. Items on the questionnaire were reversely scored and linearly transformed to a 0-100 scale, so that higher scores indicated better patient reported outcome. The mean was computed as the sum of the items over the number of items answered (to account for missing data). If more than 50% of the items in the scale were missing, the score was not computed.
Time Frame: Month 6
Population: Pediatric patients who completed the questionnaire. Because the study was terminated early with a limited number of subjects and subject visits, the data are only summarized. Too few data are available for meaningful analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open-label Herold Regimen | Double-blind Herold Regimen | Double-blind 33.3% Herold Regimen | Double-blind Curtailed Herold Regimen | Double-blind Placebo
Number analyzed (Participants) | 26 | 18 | 10 | 10 | 10
units on a scale | 7.7 (6.82) | 13.5 (13.07) | 12.2 (8.82) | 9.3 (10.52) | 13.8 (15.66)

14. Secondary Outcome: Pediatric Quality of Life Questionnaire Total Score
Description: as for outcome 13
Time Frame: Month 12
Population: Pediatric patients completing PedQL questionnaire. Because the study was terminated early with a limited number of subjects and subject visits, the data are only summarized. Too few data are available for meaningful analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open-label Herold Regimen | Double-blind Herold Regimen | Double-blind 33.3% Herold Regimen | Double-blind Curtailed Herold Regimen | Double-blind Placebo
Number analyzed (Participants) | 27 | 2 | 2 | 2 | 2
units on a scale | 6.3 (6.39) | 21.0 (26.87) | 6.5 (2.12) | 11.0 (9.90) | 30.5 (7.78)

15. Secondary Outcome: Percentage of Cells by Immunophenotype
Time Frame: Month 6
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Open-label Herold Regimen | Double-blind Herold Regimen | Double-blind 33.3% Herold Regimen | Double-blind Curtailed Herold Regimen | Double-blind Placebo
Number analyzed (Participants) | 9 | 5 | 4 | 6 | 3
Percent
  %CD25+/FOXp3+ [of CD4+] | 0.4 (1.87) | 5.5 (1.35) | 4.8 (1.00) | 6.0 (1.28) | 4.5 (1.46)
  %CD25+/FOXp3+ [of CD8+] | 0.2 (0.33) | 0.5 (0.3) | 0.4 (0.10) | 0.7 (0.46) | 0.6 (0.35)
  %CD3+/CD16,CD56+ | 6.7 (4.39) | 4.4 (1.52) | 7.7 (2.85) | 4.8 (1.63) | 4.2 (1.02)
  %CD3-/CD16,CD56+ | 8.9 (3.32) | 9.1 (3.23) | 6.4 (3.09) | 10.7 (4.31) | 5.8 (2.11)
  %CD40+ [of CD4+] | 0.7 (0.49) | 1.1 (0.48) | 0.9 (0.89) | 0.8 (0.54) | 0.8 (0.52)
  %CD69+ [of CD4+] | 0.9 (0.77) | 0.1 (0.09) | 0.7 (1.20) | 0.1 (0.12) | 0.1 (0.10)
  %CD69+ [of CD8+] | 3.7 (1.71) | 3.3 (0.23) | 3.4 (1.39) | 3.4 (1.25) | 4.2 (1.16)

16. Secondary Outcome: Human Anti-human Antibody (HAHA) Levels
Description: Patients with HAHA levels > 0.
Time Frame: Month 6 and 12
Measure: Count of Participants; unit: Participants
Arm/Group | Open-label Herold Regimen | Double-blind Herold Regimen | Double-blind 33.3% Herold Regimen | Double-blind Curtailed Herold Regimen | Double-blind Placebo
Number analyzed (Participants) | 32 | 73 | 38 | 38 | 38
Participants
  Month 6 | 30 | 22 | 13 | 12 | 11
  Month 12 | 26 | 2 | 2 | 2 | 2

ADVERSE EVENTS:
Time Frame: Throughout the study, up to 15 months
Description: Only serious adverse events and adverse events of special interest (AESI) were collected and reported in this study. AESI include non-serious infections, lymphomas or other cancers, new onset autoimmune diseases, events related to complication of diabetes, and clinically significant low blood sugar episodes requiring assistance from another individual.
Arm/Group | Open-label Herold Regimen | Double-blind Herold Regimen | Double-blind 33.3% Herold Regimen | Double-blind Curtailed Herold Regimen | Double-blind Placebo
All-Cause Mortality (participants affected / at risk) | 0/32 | 1/73 | 0/38 | 0/38 | 0/38
Serious Adverse Events (participants affected / at risk) | 1/32 | 5/73 | 3/38 | 4/38 | 0/38
Other Adverse Events (participants affected / at risk) | 8/32 | 2/73 | 1/38 | 10/38 | 4/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label Herold Regimen (N=32) | Double-blind Herold Regimen (N=73) | Double-blind 33.3% Herold Regimen (N=38) | Double-blind Curtailed Herold Regimen (N=38) | Double-blind Placebo (N=38)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 1 | 1 | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypoglycaemic seizure (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Appendicitis perforated (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Varicella (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Peritonitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Caustic injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Iritis (Eye disorders) | 0 | 0 | 0 | 1 | 0
Death (General disorders) | 0 | 1 | 0 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label Herold Regimen (N=32) | Double-blind Herold Regimen (N=73) | Double-blind 33.3% Herold Regimen (N=38) | Double-blind Curtailed Herold Regimen (N=38) | Double-blind Placebo (N=38)
Fungal skin infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Epstein-Barr virus antibody positive (Investigations) | 1 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 1 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Tinea infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Diabetic neuropathy (Nervous system disorders) | 0 | 0 | 0 | 2 | 0
Diabetic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 1 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Diabetic nephropathy (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1

LIMITATIONS AND CAVEATS:
No formal inferential analyses were conducted due to limited number of participants. Data are summarized as mean change from baseline, both from Protégé and Extension baselines, for C-peptide AUC, HbA1c, insulin, and fasting C-peptide. Only existing data are summarized, no last observation carried forward imputation was performed. Patient reported outcomes were collected and summarized as mean change from baseline. However, only change from baseline from Extension could be summarized.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes